CLINICAL TRIAL: NCT07095400
Title: Evaluation of Functional and Biochemical Effectiveness of a Strength Training Protocol in Parkinson's Disease
Acronym: POWER-PD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Villanueva (Other)
Responsible Party: Principal Investigator, Noelia Diaz Lopez, Doctor, Universidad Villanueva
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 240320252802025
Record Dates: First submitted 2025-07-21; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Parkinson Disease
Keywords: strength training; physical exercise; oxidative stress; neurofilament light chain; parkinson's disease
MeSH Terms: conditions — Parkinson Disease; Motor Activity; Charcot-Marie-Tooth disease, Type 1F | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Strength training group (Experimental): An intervention based on the application of a strength training protocol for multi-joint and single-joint muscles will be implemented, performed with a slow-moderate execution speed. This intervention will be carried out over 12 weeks, with a total of 24 sessions (2 sessions per week), each lasting 45 minutes. In all of these sessions, free weights will be used, performing three sets at 60-80% of 1RM for 8-12 repetitions.
  The exercise protocol will include:
  * Squats
  * Deadlifts
  * Rows
  * Bicep curls
  * Bench press
  * Shoulder press
  Each set will be performed to muscular failure, progressing in the number of repetitions (from 8 to 12). Once 12 repetitions are reached, the load volume will be increased by adding 5% to the weight.
  Interventions: Other: strength training

INTERVENTIONS:
Other: strength training — An intervention based on the application of a strength training protocol for multi-joint and single-joint muscles will be implemented, performed with a slow-moderate execution speed. This intervention will be carried out over 12 weeks, with a total of 24 sessions (2 sessions per week), each lasting 45 minutes. In all of these sessions, free weights will be used, performing three sets at 60-80% of 1RM for 8-12 repetitions.
  The exercise protocol will include:
  * Squats
  * Deadlifts
  * Rows
  * Bicep curls
  * Bench press
  * Shoulder press
  Each set will be performed to muscular failure, progressing in the number of repetitions (from 8 to 12). Once 12 repetitions are reached, the load volume will be increased by adding 5% to the weight.

SUMMARY:
Parkinson's Disease (PD) is a complex neurodegenerative disorder characterized by the progressive loss of dopaminergic neurons, which results in a range of motor symptoms such as tremor, rigidity, and bradykinesia, as well as non-motor symptoms including anxiety, depression, and cognitive decline. Strength training has emerged as a promising intervention to improve motor function and influence biochemical markers associated with oxidative stress and neurodegeneration. This study aims to evaluate the effectiveness of a structured strength training protocol over 12 weeks in improving both functional and biochemical outcomes in patients with PD.

DETAILED DESCRIPTION:
Parkinson's Disease (PD) is a multifaceted neurodegenerative condition marked by the gradual degeneration of dopaminergic neurons, causing a spectrum of motor impairments-such as tremor, rigidity, and bradykinesia-and non-motor challenges, including anxiety, depression, and cognitive decline. Previous research indicates that strength training can positively impact both the motor abilities and certain biochemical parameters related to oxidative stress and neurodegeneration in individuals with PD.

This study is designed as a quasi-experimental, prospective, longitudinal investigation involving patients recruited from a specialized care center for PD. Over the course of 12 weeks, participants will engage in a strength training program consisting of 24 sessions (twice weekly). The primary objective is to assess changes in functional outcomes and biochemical markers, with secondary aims addressing balance, gait, psychological status, cognitive function, and overall quality of life.

Functional assessments will include tests such as the Timed Up and Go Test, Berg Balance Scale, 10-Meter Walk Test, and the 30-Second Sit-to-Stand Test. Cognitive and emotional functions will be evaluated using the Mini-Mental State Examination, GAD-7, and PHQ-9 questionnaires, while quality of life will be measured with the PDQ-39 questionnaire. Biochemical analyses will focus on markers of oxidative stress-Malondialdehyde (MDA), 8-OHdG, Total Antioxidant Capacity (TAC)-and neurodegeneration via neurofilament light chain (NfL) levels.

Through this comprehensive approach, the study seeks to contribute valuable evidence on the benefits of strength training in PD and aims to optimize therapeutic protocols that enhance the quality of life and functional independence of affected patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with PD who meet the modified diagnostic criteria of the UK Brain Bank.
* Patients in stage II or III of the Hoehn and Yahr Scale.
* A score greater than 60% on the Schwab and England Functional Scale.
* Patients whose motor response to pharmacological treatment is stable or slightly fluctuating and who are not receiving any specific strength training rehabilitation treatment at the time of the study.

Exclusion Criteria:

* Diagnosis of a condition other than PD.
* Significant comorbidities and/or severe systemic diseases that would prevent participation in exercise (e.g., recent surgery, cardiac instability, anemia, hepatosis, pulmonary disorders, chronic renal failure, or severe mental disorders).
* Inability to actively understand instructions and cooperate in the tasks given, based on a score <24 on the Mini-Mental State Examination (MMSE).
* Refusal to participate in the study.
* Stages I, IV, or V of the Hoehn and Yahr Scale.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2025-09-07 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Timed Up and Go Test | 12 weeks
  Test developed to evaluate balance and functional mobility to determine the risk of falling. The test consists of timing how long it takes the subject to perform the action of standing up from a chair, walking 3 meters in a straight line, turning around, and sitting back down in the chair. An increase in the time taken to complete the test indicates worse outcomes.
Berg Balance Scale | 12 weeks
  Scale developed to evaluate balance and postural control. The scale consists of 14 items with Likert-type responses ranging from 0 to 4, where 0 represents the lowest level of function and 4 represents the highest level of function. Higher values indicate better balance control.
10 meter walk test | 12 weeks
  Instrument used to evaluate gait speed in meters per second. The test consists of timing how long it takes the subject to cover a 10-meter straight path (to avoid acceleration-deceleration effects, 2 meters are added at the beginning and end of the path). An increase in the time taken to complete the test indicates worse outcomes.
30 second sit to stand test | 12 weeks
  Instrument used to evaluate the strength and endurance of the lower limbs. The test is performed with a 43 cm chair without armrests; the number of squats the subject is able to perform in 30 seconds is counted. The higher the number of squats performed, the better the test results.
Parkinson's Disease Questionnaire (PDQ-39) | 12 weeks
  It is an instrument that evaluates the quality of life in patients with Parkinson's disease. It includes 8 areas: mobility, activities of daily living, emotional well-being, stigma, social support, cognition, communication, and bodily discomfort. Higher scores on the PDQ-39-SV scale indicate worse outcomes.
Mini-Mental State Examination | 12 weeks
  It is a widely used screening tool for assessing cognitive function. It is commonly employed to detect cognitive impairment and monitor changes over time in conditions such as dementia or following neurological events like stroke or traumatic brain injury. The total score ranges from 0 to 30. A higher score indicates better cognitive performance and less impairment.
Patient Health Questionnaire-9 (PHQ-9) | 12 weeks
  It is an instrument that assesses the severity of depressive symptoms. The total score range from 0 to 27. Each of the nine items is rated on a scale from 0 to 3, resulting in a minimum score of 0 (indicating no depressive symptoms) and a maximum score of 27 (indicating severe depression). Higher scores indicate greater severity of depressive symptoms.
Malondialdehyde (MDA) | 12 weeks
  MDA, measured in nanomoles per milliliter (nmol/mL), is a byproduct of lipid peroxidation and one of the most widely studied markers of oxidative tissue damage, particularly during exercise.
  Higher MDA levels indicate greater lipid oxidative damage, suggesting a more harmful oxidative environment. MDA levels will be assessed using ELISA according to the manufacturer's instructions.
8-Hydroxy-2'-deoxyguanosine (8-OHdG) | 12 weeks
  8-OHdG is a marker of oxidative damage to DNA, typically measured in nanograms per milliliter (ng/mL) or nanomoles per liter (nmol/L).
  Elevated 8-OHdG levels reflect increased DNA oxidation, which is associated with cellular aging and neurodegenerative processes. Quantification will be performed using ELISA, following the manufacturer's protocol.
Total Antioxidant Capacity (TAC) | 12 weeks
  TAC reflects the overall antioxidant defense and is generally expressed in millimoles of Trolox equivalents per liter (mmol Trolox/L).
  Higher TAC values indicate stronger antioxidant capacity, suggesting a more favorable redox balance. TAC will be analyzed using ELISA in accordance with the manufacturer's instructions.
Neurofilament Light Chain (NfL) | 12 weeks
  NfL, measured in picograms per milliliter (pg/mL), is a well-established biomarker of neuroaxonal damage and neurodegeneration, released into extracellular fluids following axonal injury.
  Higher NfL levels indicate greater neuroaxonal damage, and thus worse neurological status. Levels of NfL will be determined using ELISA, following the manufacturer's recommendations.

CONTACTS AND LOCATIONS:
Overall Officials: Noelia Díaz López, Doctor, Study Director — Universidad Villanueva
Locations (1):
- Universidad Villanueva, Madrid, Madrid, Spain